CLINICAL TRIAL: NCT04138186
Title: A Randomized, Placebo Controlled, Double-blind, Parallel-arm Feasibility (Pilot) Study to Evaluate Safety and Clinical Efficacy of G-PUR® Treatment in Patients With Irritable Bowel Syndrome With Diarrhea (IBS-D)
Brief Title: G-PUR® for Symptomatic Treatment in Irritable Bowel Syndrome With Diarrhea
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Glock Health, Science and Research GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: G-IBS_01
Record Dates: First submitted 2019-10-16; First posted 2019-10-24 (Actual); Last update posted 2020-11-13 (Actual); Status verified 2020-11

CONDITIONS: Irritable Bowel Syndrome With Diarrhea (IBS-D)
Keywords: IBS; Diarrhea; Gastrointestinal function disorder
MeSH Terms: conditions — Diarrhea | interventions — Administration, Oral

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 2.0g G-PUR® capsules (Experimental)
  Interventions: Device: 2.0g G-PUR®, oral administration
- Placebo capsules (Placebo Comparator)
  Interventions: Device: Placebo, oral administration

INTERVENTIONS:
Device: 2.0g G-PUR®, oral administration — tid for 12 weeks
  Arms: 2.0g G-PUR® capsules
Device: Placebo, oral administration — tid for 12 weeks
  Arms: Placebo capsules

SUMMARY:
A randomized, double-blind, placebo-controlled pilot study in patients with IBS-D according to Rome IV criteria evaluating the clinical efficacy and safety of oral administration of 2g G-PUR® tid compared to placebo in a cohort of 30 patients over an active treatment period of 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-75 years
2. Recurrent abdominal pain, at least one day/week in the last 3 months (with symptom onset at least 6 months before diagnosis), associated with two or more of the following criteria (Rome IV criteria)

   1. Related to defecation
   2. Associated with a change in frequency of stool
   3. Associated with a change in form (appearance) of stool.
3. Moderate to severe abdominal pain as defined with an IBS Symptoms Severity Scale (IBS-SSS) score > 175
4. Patient reports that abnormal bowel movements are usually diarrhea with more than one-fourth (25%) of bowel movements with Bristol stool form types 6 or 7 and less than one-fourth (25%) of bowel movements with Bristol stool form types 1 or 2. Starting during the screening/run-in phase, all patients will keep diaries of stool frequency and consistency. Stool consistency will be assessed according to the Bristol Stool Form scale (Lewis and Heaton, 1997)
5. Stable eating habits, within one month before randomization
6. In patients > 50 years colonoscopy performed during the past 5 years demonstrates no pathology associated with the symptoms reported for IBS
7. Ability to understand trial instructions and to comply with treatment
8. Patient agree to be compliant for study interactive web - response system schedule confirmed at time of randomization
9. Written informed consent prior to enrolment

Exclusion Criteria:

1. Patient has exclusively constipation-predominant IBS (IBS-C) that is characterized by < 3 bowel movements/week or hard and lumpy stools (e.g. Bristol stool form types 1 or 2)
2. Patient has irritable bowel syndrome with mixed bowel habits (IBS-M) with varying symptoms of constipation and diarrhea
3. Calprotectin stool value > 200mg/kg stool
4. Known hypersensitivity to the IMD (known aluminium and/or silicon hypersensitivity)
5. Patient has failed to record >50% of daily diary entries during run-in period
6. Rectal bleeding in the absence of documented bleeding hemorrhoids or anal fissures assessed by fecal occult blood test
7. History of major gastric, hepatic, pancreatic or intestinal surgery or perforation with exception of appendectomy, cholecystectomy and inguinal hernia
8. Patients with a history of positive tests for ova, parasites or clostridium difficile must undergo repeat testing, which must be negative, during the screening period
9. Use of the following prohibited medications: any antibiotics including rifaximin within the past 2 months or during treatment period, use of cholestyramine during entire study period, during run-in phase and during the treatment period any use of concomitant medication effecting the gastrointestinal movement and/or function (e.g. anticholinergic drugs, 5-HT3 receptor antagonists, prokinetic agents, intestinal flora regulating drugs, parasympathetic inhibitors, opioids or eluxadoline)
10. Use of immunosuppressive drugs within the last 6 months or planned use of immunosuppressive drugs during the study
11. Patients treated with tricyclic antidepressants
12. Serotonin re-uptake inhibitors are allowed if the patient is at stable dose for at least 8 weeks prior to signing informed consent and the dose will remain stable throughout the duration of the study.
13. History of inflammatory or immune-mediated gastrointestinal (GI) disorders including inflammatory bowel disease (i.e., Crohn's disease, ulcerative colitis) and celiac disease (by anamnesis and assessed by tTGA levels)
14. Active infection, or abnormalities in laboratory testing, vital signs, or physical examination at screening
15. Participation in any other interventional clinical trial within 4 weeks before study participation
16. Alcohol or drug abuse (History of alcohol abuse or heavy alcohol use as binge drinking on 5 or more days per month within the 12 months prior to screening. Known medication and drug abuse)
17. Pregnant or breastfeeding (for all females, negative pregnancy test at screening and at each treatment visit will be performed).
18. History of cancer (except non-melanoma skin cancer, or carcinoma in situ of cervix) within the previous 12 months or treatment with anticancer therapy (chemotherapy, immunotherapy, radiotherapy, hormone therapy for cancer treatment, targeted therapy or gene therapy) within 12 months before the first administration of investigational product or at any time during the study
19. Patients with known familial colorectal cancer syndromes, where colorectal cancer has not been excluded by colonoscopy
20. Other severe comorbid condition, concurrent medication, or other issue that renders the patient unsuitable for participation in the study, including but not limited to: comorbid condition with an estimated life expectancy of ≤ 12 months, patients with uncontrolled hypothyroidism, uncontrolled hyperthyroidism, patients on dialysis, patients with severe pulmonary (requiring home oxygen, uncontrolled COPD Gold III/ IV) or cardiovascular conditions (heart failure NYHA III and IV, uncontrolled hypertension systolic BP by repeated measurement > 180 mmHg; patient with uncontrolled diabetes with an Hba1c >6.5%)
21. Concomitant psychotherapy is allowed if the patient started therapy for at least 8 weeks prior to signing informed consent and the schedule will remain stable throughout the duration of the study.
22. Known severe psychiatric disorders or mental condition rendering the patient unable to understand the nature, scope and possible consequences of the study;
23. Presence of any condition that impacts compliance with the study procedures
24. Employee at the study site, spouse/partner or relative of any study staff (e.g. investigator, sub-investigators, or study nurse) or relationship to the sponsor)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-10-02 (Actual); Primary Completion 2021-02 (Estimated); Study Completion 2021-02 (Estimated)

PRIMARY OUTCOMES:
The rate of responders for the patient's global assessment of relief using the last four assessments in the treatment period. | 12 weeks

SECONDARY OUTCOMES:
Patient's global assessment of symptom relief measured on a 5-point Likert scale (1= very good and 5= very poor) | 12 weeks
Incidence of adverse (and serious) events | 12 weeks
Daily intensity of bloating using a 11-point numerical rating scale (NRS) where 0 represents no bloating discomfort and 10 represents very severe bloating discomfort | 12 weeks
Daily urgency using a 11-point numerical rating scale (NRS) where 0 represents no defecation urgency and 10 represents worst imaginable urgency | 12 weeks
Daily stool frequency | 12 weeks
  Daily Stool Frequency assessed by daily diary entry of the total number of bowel movements within the last 24 hours
Patient compliance with daily diary reporting | 12 weeks
ePRO usability using a paper questionnaire | 12 weeks
Worst daily abdominal pain using a 11-point NRS | 12 weeks
  Percentage of responders, defined as the percentage of participants who meet the following criterion for at least 50% of the days with diary entry: Abdominal pain assessed by a 11-point NRS-scale improved at least 30% compared to baseline
Daily stool consistency using the Bristol Stool Form Scale (Type 1 separate hard lumps, like nuts (hard to pass); Type 7 watery, no solid pieces, entirely liquid) | 12 weeks
  Percentage of responders, defined as the percentage of participants who have ≥50% reduction in the number of days per week with at least one stool that has a consistency of Type 6 or 7 on the Bristol stool scale compared to baseline
Responder rate (ie weekly and daily) of the combined endpoint: worst daily abdominal pain and daily stool consistency | 12 weeks
Additional responder analyses (i.e. weekly and daily) of IBS symptoms listed all above evaluating different change in symptom intensity with treatment (i.e., greater than or equal to 30, 40 and 50 percent change in intensity compared with baseline) | 12 weeks
Number of pain-free days | 12 weeks
Assessment of gastrointestinal symptoms using the IBS-SSS during each onsite visit; | 12 weeks
  Proportion of patients having a reduction ≥ 50 on the IBS-SSS system (ranges 0-500). A decrease in 50 or greater in the IBS-SSS is considered a positive response.
Quality of Life using validated generic SF12 questionnaire | 12 weeks
Hospital anxiety and depression scale (HADS) | 12 weeks
  scale measuring anxiety and depression (14 items); likert scale 0 (not at all) to 3 (most of the time); higher scores(summed) indicate presence of anxiety or depression
Stress response using the perceived stress questionnaire | 12 weeks
  The (Perceived Stress Questionnaire) PSQ consists of 30 items, each of which has to be scored by a test person using a Likert scale (1 for "almost never", 2 for "sometimes", 3 for "frequently" to 4 for "mostly") how often each item/sentence applied during the last month. Each number has a point that reveals the level of stress for each sentence. Points are calculated according to the calculation system of the scale, and for each individual, the final calculation results in the total value between 0 and 100. Higher total values indicate more stress
Use of rescue medication (to be assessed daily) | 12 weeks
Exploratory endpoint: bile acid in stool | 12 weeks
  bile acid excretion in stool before and after 12 weeks treatment
Exploratory endpoint: zonulin in stool | 12 weeks
  zonulin (ng/ml) in stool before and after 12 weeks treatment
Exploratory endpoint: microbiome in stool | 12 weeks
  microbiome in stool assessed by 16S gene sequencing before and after 12 weeks treatment
Exploratory endpoint: HBD2 in stool | 12 weeks
  human beta defensin 2 (HBD2) (ng/ml) in stool before and after 12 weeks treatment
Exploratory endpoint: gluten in stool | 12 weeks
  gluten (ng/ml) in stool before and after 12 weeks treatment
Exploratory endpoint: IDO in blood | 12 weeks
  indoleamine-2,3- dioxygenase (IDO) (umol/mmol) in capillary blood before and after 12 weeks treatment
Exploratory endpoint: zonulin in blood | 12 weeks
  zonulin (ng/ml) in capillary blood before and after 12 weeks treatment

CONTACTS AND LOCATIONS:
Overall Officials: Michael Wolzt, Prof. Dr., Principal Investigator — Department of Clinical Pharmacology, Medical University of Vienna
Locations (1):
- Department of Clinical Pharmacology, Medical University of Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No